CLINICAL TRIAL: NCT03473483
Title: Cigarette Harm Reduction With Electronic Cigarette Use
Acronym: NIDA-SREC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Major study re-design prior to participant enrollment
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 17-23142; U01DA045519 (NIH)
Record Dates: First submitted 2018-02-09; First posted 2018-03-22 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Nicotine Dependence; Tobacco Toxicity; Nicotine Dependence, Cigarettes; Cardiovascular Risk Factor; Nicotine Withdrawal
Keywords: nicotine; tobacco; research electronic cigarette; e-cigarette; SREC
MeSH Terms: conditions — Tobacco Use Disorder; Vaping

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SREC only or cigarette only use (Experimental): Four days of SREC/Usual cigarette/product use as regular with daily diary. Admitted to hospital research ward on Day 5 and 6 for 2 hospital day visits that includes a standardized session of product use; 4-hr abstinence; pharmacokinetic (PK) blood draws; ad libitum use of product; cardiovascular (CV) monitoring, 12-hr urine collections, and 12-hr circadian blood draws.
  Interventions: Other: SREC
- Alternate product from Arm 1 (Experimental): Four days of SREC/Usual cigarette/product use as regular with daily diary. Admitted to hospital research ward on Day 5 and 6 for 2 hospital day visits that includes a standardized session of product use; 4-hr abstinence; PK blood draws; ad libitum use of product; CV monitoring, 12-hr urine collections, and 12-hr circadian blood draws.
  Interventions: Other: SREC
- Standardized Dual Use (Experimental): Four days of SREC and/or usual product use as regular with daily diary. Admitted to hospital research ward on Day 5 and 6 for 2 hospital day visits that includes ad libitum SREC use and less than usual amount of cigarette use; CV monitoring, 12-hr urine collections, and 12-hr circadian blood draws.
  Interventions: Other: SREC

INTERVENTIONS:
Other: SREC — The Standardized Research E-Cigarette (SREC) was developed by NIDA to help researchers assess uncertainties in electronic nicotine delivery devices.
  Tank:
  * Sealed and disposable
  * Minimum 350 puffs per tank
  * Volume of e-liquid per tank ~ 3ml
  E-Liquid Characteristics:
  * Tobacco flavored
  * Nicotine concentration: 15 mg/ml
  * Propylene Glycol:~ 50% (wt / wt)
  * Glycerin: ~ 50% (wt / wt)
  * Cotinine: <1 μg/g
  * Nornicotine: 5 μg/g
  * Myosmine : 3 μg/g
  * Anabasine: <1 μg/g
  * Anatabine: <1 μg/g
  * Beta:nicotyrine: <1 μg/g
  * Diacetyl: <2 μg/g
  * 2,3:Pentanedione: <1 μg/g
  * Arsenic: <0.1 μg/g
  * Cadmium: <0.1 μg/g
  * Chromium: <0.1 μg/g
  * Lead: <0.1 μg/g
  * Nickel: <0.1 μg/g
  * Mercury: <0.05 μg/g
  Other Names: Standardized Research E-Cigarette

SUMMARY:
This is an observational, crossover study that will be examine use behaviors, chemical exposures, and biological effects of SREC compared to TC use in subjects confined to a research ward setting.

DETAILED DESCRIPTION:
Daily cigarette smokers who are familiar with e-cigarette (EC) use will be instructed to use only NIDA Standardized Research Electronic Cigarettes (SREC) and tobacco cigarettes (TC) while enrolled on the study. Our overall goals are two-fold: (1) to compare nicotine and toxicant exposure and pharmacological effects of SREC used alone vs tobacco cigarettes alone (TC), or dual use; and (2) using SREC alone, TC alone, or ad libitum SREC use combined with 50% reduction in usual TC use as a model for dual use, to examine the extent to which nicotine and toxicant exposure and biomarkers of potential harm compare among the 3 groups. The former would inform the effects of total switching, the latter would inform the potential harm reducing effects of smoking fewer TC while using EC.

ELIGIBILITY:
Inclusion Criteria:

* Healthy on the basis of medical history and limited physical examination as described below:
* - Heart rate < 105 beats per minute (BPM)
* - Systolic Blood Pressure < 160 and > 90
* - Diastolic Blood Pressure < 100 and > 50
* - Body Mass Index ≤ 38.0
* - Expired Carbon Dioxide (CO) >=5ppm
* Current regular "dual" user of both electronic cigarette (EC) and tobacco cigarette (TC)
* EC device use at least 10 or more days in the past 30 days
* Daily use of conventional TC (at least 10 cigarettes per day (CPD), as confirmed by saliva cotinine >50 ng/ml and/or NicAlert=6)
* Age: >= 21 years old to <= 70 years old
* Willingness to use a non-menthol e-cigarette only (until menthol flavored SREC becomes available)
* Willingness to abstain from marijuana for the duration of the study

Exclusion Criteria:

* Unstable medical conditions (such as unstable heart disease, seizures, cancer, uncontrolled thyroid disease, diabetes, Hepatitis B or C or renal or liver impairment, glaucoma, history of stroke, an ulcer in the past year, or active use of an inhaler for Asthma or Chronic obstructive pulmonary disease (COPD).
* Psychiatric conditions (such as current or past schizophrenia and/or current or past bipolar disorder, major personality disorder, or major depression current or within the past year. Participants with current or past minor to moderate depression and/or anxiety disorders will be reviewed by the study physician and considered for inclusion. Psychiatric hospitalizations are not exclusionary, but study participation will be determined as per study physician's approval.
* Psychiatric medications with the exception of Selective Serotonin Reuptake Inhibitors (SSRI) and Serotonin and norepinephrine reuptake inhibitors (SNRIs) and current evaluation by the study physician that the participant is otherwise healthy, stable and able to participate.
* Pregnancy or breastfeeding (by history and pregnancy test); women of childbearing potential must be using an acceptable method of contraception
* Concurrent regular use of marijuana [occasional users of these products may be enrolled if they agree to abstain from their use during the period of the study]
* Use of other tobacco products, smokeless tobacco, pipes, cigars/cigarillos, blunts/spliffs [no more than 15 times in combination in the past month and must agree to abstain from their use during the period of the study.]
* Concurrent use of nicotine-containing medications
* Alcohol or illicit drug dependence within the past 12 months (with the exception of those who have recently completed an alcohol/drug treatment program). Positive toxicology test at the screening visit (THC ok). Must not be on opioid replacement therapy.
* Medications: Use of medications that are inducers of nicotine metabolizing enzyme CYP2A6 (Example: rifampicin, dexamethasone, phenobarbital, and other anticonvulsant drugs). Use of medications for cardiovascular conditions including hypertension (Example: beta- and alpha-blocking drugs). Use of stimulants (Example: Adderall)
* Other/Misc Health Conditions: Oral thrush; fainting within the last 30 days; untreated thyroid disease; other "life threatening illnesses" as per study physician's discretion.
* Concurrent participation in another clinical trial
* Inability to read and write in English
* Planning to quit smoking or vaping within the next 60 days
* A known propylene glycol/vegetable glycerin allergy

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Peak Nicotine Concentration | Up to 2 years
  Compare peak nicotine concentration between SREC vs. Tobacco Cigarette (TC) use
Time of Peak Nicotine Concentration | Up to 2 years
  Compare time of peak nicotine concentration between SREC vs. Tobacco Cigarette (TC) use
Mean overall systemic nicotine exposure | Baseline through study completion, approximately 2 years
  Descriptive statistics will be used to examine systemic nicotine exposure from daily use of SREC and compare daily nicotine intake to TC use
Change in Mean score on the Modified Cigarette Evaluation Questionnaire (mCEQ) | Baseline through study completion, approximately 2 years
  The mCEQ use three multi-item domains (subscales) and two single items: "Smoking Satisfaction", "Psychological Reward", "Aversion", "Enjoyment of Respiratory Tract Sensations" and "Craving Reduction". Scores for each subscale are calculated as the average of its individual item responses of The items are rated on a seven-point scale ranging from 1 (not at all) to 7 (extremely). Higher scores indicate greater intensity of each smoking effect with, for example, greater satisfaction or psychological reward after smoking. Scores will be compared between SREC, TC, and dual use
Patterns of puffing | Baseline through study completion, approximately 2 years
  Compare the pattern of puffing between SREC and TC use by coding the recorded ad libitum use of SREC vs TC.
Change in Mean score on the Minnesota Tobacco Withdrawal Scale-Revised (MTWS-R) | Baseline through study completion, approximately 2 years
  The MTWS-R features two separate measures for examining the severity of nicotine withdrawal symptoms in a participant: a self-report scale and an observer scale. The observer scale asks the scale-taker to rate the severity of four symptoms in someone the they know who is experiencing nicotine withdrawal: "angry/irritable/frustrated," "anxious/tense," "depressed," and "restless/impatient." The self-report version asks for rankings of the severity of those same four symptoms, plus eleven others that cannot be observed by outsiders (including such things as "desire or craving to smoke," "insomnia, sleep problems, awakening at night," or "dizziness). Both scales use a Likert-type scale for the severity ratings, ranging from 0 ("not at all") to 4 ("severe"). These scores are tallied to calculate an a total withdrawal discomfort score and will be compared between SREC, TC, and dual use.
Change in Mean score on the Questionnaire on Smoking Urges (QSU-Brief) | Baseline through study completion, approximately 2 years
  The QSU-Brief consists of 10 statements about the respondent's feelings and thoughts about his or her desire to smoke cigarettes as he or she is completing the questionnaire (i.e., right now). Each response is scored a number ranging from 1 (strongly disagree) to 7 (strongly agree) and total scores are calculated by summing the item scores to compare craving between SREC, TC, and dual use.
Change in Mean score on the Positive and Negative Affect Scale (PANAS) | Baseline through study completion, approximately 2 years
  The Positive and Negative Affect Schedule (PANAS) is a brief scale is comprised of 20 items, with 10 items measuring positive affect (e.g., excited, inspired) and 10 items measuring negative affect (e.g., upset, afraid). Each item is rated on a five-point Likert Scale, ranging from 1 = Very Slightly or Not at all to 5 = Extremely, to measure the extent to which the affect has been experienced in a specified time frame and the final score is derived out of the sum of the ten items on both the positive and negative side. Scores can range from 10-50 for both the Positive and Negative Affect with the lower scores representing lower levels of Positive/Negative Affect and higher scores representing higher levels of Positive/Negative Affect. The scores will be comparted between SREC, TC, and dual use.

SECONDARY OUTCOMES:
Changes in mean circadian heart rate | Baseline through study completion, approximately 2 years
  Compare changes in mean circadian heart rate between SREC-only and TC-only use
Changes in mean blood pressure | Baseline through study completion, approximately 2 years
  Compare changes in blood pressure between SREC-only and TC-only use
Changes in mean urinary catecholamine | Baseline through study completion, approximately 2 years
  Compare mean urinary catecholamine excretion between SREC-only and TC-only use
Mean Level of exposure to Tobacco smoke toxicant | Baseline through study completion, approximately 2 years
  Compare levels of exposure of tobacco smoke toxicant between dual SREC-TC use and TC-only use
Sensitivity of anabasine or nicotelline to nicotine metabolites | Baseline through study completion, approximately 2 years
  Sensitivity is defined as the ratio of anabasine or nicotelline to nicotine metabolites (cotinine or total nicotine equivalents) in urine from SREC-only and TC-only use.
Specificity of anabasine or nicotelline to nicotine metabolites | Baseline through study completion, approximately 2 years
  Specificity of anabasine or nicotelline will be compared to nicotine metabolites (cotinine or total nicotine equivalents) in urine from SREC-only and TC-only use.

CONTACTS AND LOCATIONS:
Overall Officials: Neal L. Benowitz, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Tobacco Research Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-11-30): https://cdn.clinicaltrials.gov/large-docs/83/NCT03473483/Prot_SAP_ICF_001.pdf